CLINICAL TRIAL: NCT04874064
Title: Triple Negative Breast Cancer Markers in Liquid Biopsies Using Artificial Intelligence (TRICIA Study)
Brief Title: TRIple Negative Breast Cancer Markers In Liquid Biopsies Using Artificial Intelligence
Acronym: TRICIA
Status: Recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Collaborators: Exactis Innovation (Other)
Responsible Party: Principal Investigator, Mark Basik, Breast Surgeon, Jewish General Hospital
Other Study IDs: TRICIA
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Liquid Biopsy; Artificial Intelligence
MeSH Terms: conditions — Breast Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood sample DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Liquid Biopsy — Blood collection and access to residual tumor.

SUMMARY:
Triple negative breast cancer (TNBC) is the most aggressive of breast cancers and it is usually treated with chemotherapy even before surgery. In many cases, the chemotherapy completely "melts" the tumor and these patients do well. When the tumor is not eliminated by the chemotherapy, the patient receive more chemotherapy after surgery to decrease the chances of it coming back. Yet many of these patients don't need that extra chemotherapy and will do well in any case. One of the most exciting recent developments in cancer is the use of "liquid biopsies". It turns out that the tumor's DNA, RNA and proteins can be detected in small vesicles found in the patient's blood. Thanks to advances in Artificial Intelligence, there is now informatics tools to integrate many types of molecular information. Our industrial partner, MIMs, will apply novel informatics tools to generate a test using all the molecular information obtained from blood vesicles and tissue that will be able to find out early if tumor has spread outside of the breast, and how much tumor is left after surgery. The goal is hope to develop a multi-dimensional test for TNBC patients that can be used to decide how much treatment they need and if treatment given after surgery is working.

DETAILED DESCRIPTION:
Rationale: The most aggressive form of breast cancer is triple negative breast cancer (TNBC), so called because these tumors do not express hormone receptors or HER2 receptor, and therefore have no readily targetable molecules. Chemotherapy is the only treatment, with chemoresistance signaling a very poor outcome even in early TNBC. The presence of residual tumor at surgery (non-pathological complete response or non-pCR) signals chemoresistance and poor prognosis, with about 30-40% of these patients dying of TNBC within the first 5 years after surgery. A recent clinical trial showed that the addition of further chemotherapy (Capecitabine) results in improved survival in these patients with non-pCR, although only about 15% of such patients do benefit. One of the most urgent unmet needs is to identify patients who will do well despite non-pCR (so as to avoid extra chemotherapy) and who will do poorly despite it, and also to identify factors of poor prognosis that may lead to novel therapeutic strategies in this group.

Current state of advancement of the technology: Until now, no biomarker except BRCA1/2 mutations has demonstrated clinical utility in the treatment of TNBC, likely due to the complex biology and heterogeneity of the disease. With the recent advances in Artificial Intelligence methodology, combining and integrating several layers of molecular data to predict outcome, until now challenging, becomes a reality. The hypothesize is that combining multi-dimensional data of tumor and plasma EVs can facilitate the development of prognostic and predictive signatures in this very aggressive disease.

Preliminary data: Thanks to our Q-CROC-03 biopsy driven clinical trial where tumor and plasma from patients with TNBC resistant to chemotherapy were collected. Whole exome seq data were translated to generate personalized circulating tumor DNA (ctDNA) assays. Our data shows a potential prognostic value to the detection of ctDNA after pre-operative chemotherapy. There is a collaboration established with Rodney Ouellette (ACRI) to isolate and profile extracellular vesicles (EVs) from plasma.

Objectives: The objective of the present study is to develop signatures of good and poor outcome as well of tumor response to chemotherapy in TNBCs by integrating multidimensional profiling of both tumor and liquid biopsies making use of Artificial Intelligence (AI) tools.

Experimental approach: EVs profiling from plasma collected in the Q-CROC-03 trial and the JGH biobank (prior, during and after chemotherapy treatment) will be performed. Profiling will include Whole Genome Sequencing (GWS), proteomics, transcriptomics and miRNA analysis. In collaboration with our industrial partner, My Intelligent Machines (MIMs), experts in bioinformatics and AI, machine-learning algorithms will be developed to integrate OMICs data from resistant tumors with matched plasma EVs data and generate a tumor/plasma signature associated with poor outcome. In parallel, in collaboration with the EXACTIS Innovation Network, patients recruitment, collection of residual tumors post chemotherapy and matched serial plasma samples during capecitabine treatment after surgery to perform the validation of the signature identified, the tumor/EV signature will be associated with patient survival.

Milestones of the proposed project: 1. Profiling of EVs from plasma. 2. Profiling of chemoresistant tumors 3. Development of algorithms to integrate multidimensional data from tumor and EVs.

The developed signatures will be IP protected. Academic and industrial partners will have shared IP (respective % to be determined). Prognostic tests will be developed on identified biomarkers and distributed through MIMsOmic Platform. MIMsOmic is an AI-powered platform commercialized by MIMs and enabling an easy, efficient and cost-effective delivery of clinical tests involving Omic data analysis.

The present project will develop a biomarker signature of poor prognosis for the most aggressive type of breast cancer. This signature will allow the identification of patients who should not be treated with post-surgery chemotherapy, and avoid unnecessary exposure to the toxicity associated with this drug.

ELIGIBILITY:
Inclusion Criteria:

* Triple negative (ER negative, PR negative and Her2 negative as defined by local standards). ER <10% is acceptable.
* Patients who have completed a minimum of 8 weeks of neoadjuvant chemotherapy.
* A cohort of TNBC patients who are awaiting surgery that have clinical or radiological evidence of residual tumor prior to surgery. This evaluation will be made at the discretion of the treating physician.

OR A second cohort of TNBC patients will be recruited after surgery, in which pathological evaluation has demonstrated the presence of residual tumor post-surgery.

* Patients who can come to the clinic for standard of care follow-up within 6 weeks post-surgery and in the next 6 months after surgery.
* Patients who are willing to provide serial blood samples.
* Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.

Exclusion Criteria:

* Clinical or radiological evidence of metastatic disease.
* Patient with a recurrence of breast cancer.
* Patients who have not had neoadjuvant chemotherapy or less than 8 weeks of neoadjuvant chemotherapy.
* Patient who received radiotherapy treatment prior to surgery.
* Patients who are not capable of signing or understanding the informed consent form.
* Known infection with HIV or hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in patients with a diagnosis of breast cancer and pathologically identified as triple negative (not expressing estrogen receptor (ER), progesterone receptor (PR) and HER2 protein, and not showing ERBB2 gene amplification) who will be undergoing neoadjuvant treatment and has residual tumor.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Develop signatures of good and poor outcome as well of tumor response to chemotherapy in TNBCs by integrating multidimensional profiling of both tumor and liquid biopsies making use of Artificial Intelligence (AI) tools | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Basik, Dr, Principal Investigator — Study Principal Investigator
Locations (3):
- Canada (3):
  - St. Joseph's Health Care London, London, Ontario
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No